CLINICAL TRIAL: NCT01033019
Title: Double-blind, Randomized, Vehicle-controlled Proof of Concept Study on the Efficacy, Safety, Local Tolerability, PK and Pharmacodynamics of Multiple Topical Administrations of LDE225 on Sporadic Superficial and Nodular Skin Basal Cell Carcinomas
Brief Title: To Evaluate the Safety, Local Tolerability, PK and PD of LDE225 on Sporadic Superficial and Nodular Skin Basal Cell Carcinomas (sBCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The data from participants with sBCCs showed insufficient efficacy with current formulation and treatment conditions.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLDE225B2204; 2009-013665-26; EudraCT 2009-013665-26
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Sporadic Superficial and Nodular Skin Basal Cell Carcinomas
Keywords: Basal cell carcinomas,; sporadic,; superficial and nodular,; skin
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDE225 0.75% (Experimental): Participants topically applied 0.75% LDE225 cream twice daily for 6 weeks.
  Interventions: Drug: LDE225 0.75%
- Vehicle (Placebo Comparator): Participants topically applied matching placebo cream twice daily for 6 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: LDE225 0.75% — 0.75% cream
  Arms: LDE225 0.75%
Drug: Vehicle — matching placebo cream to 0.75% LDE225 cream
  Arms: Vehicle

SUMMARY:
This was a double-blinded, randomized, vehicle-controlled study in sporadic superficial BCC (sBCC) and nodular BCC (nBCC) patients which consisted of a 21-day screening period, a treatment period of 6 weeks (topical 0.75% LDE225 cream application b.i.d) ending with post treatment biopsies, as safety visit one week after final study drug administration (Day 50), a visit on Day 83 for excision of the treated BCC, and an end of study evaluation (Day 90).

ELIGIBILITY:
Inclusion Criteria:

* Patients with one histologically confirmed superficial and nodular basal cell carcinoma (8-20 mm) eligible for surgical excision on selected body areas (scalp, arm, frontal trunk, posterior trunk, upper legs)

Exclusion Criteria:

* Previous treatment of the sBCC that are selected for treatment.
* Any systemic treatment which is known to affect BCCs esp. cytostatic treatments, retinoids and photodynamic treatments.
* Dark-skinned persons whose skin color prevents readily assessment of skin reactions

Other protocol defined Incl./Excl. criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Australia (2):
  - Novartis Investigative Site, Benowa, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna

REFERENCES:
- See also: Related Info — http://www.NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-five participants were enrolled into the trial. However, one participant was excluded from the efficacy analysis. Therefore, the enrollment number differs from the number started below.
Period: Overall Study
Arm/Group | LDE225 0.75% | Vehicle
Started | 16 | 8
Completed | 15 | 8
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LDE225 0.75% | Vehicle | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (7.3) | 63 (7.5) | 63 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Clinical Evaluation of sBCCs Tumors
Description: The clinical response parameters were defined as (i) complete response (i.e., there is no longer any visible evidence of a lesion consistent with BCC at this site), (ii) partial response (i.e., although a BCC still remains at this site, it has demonstrated a visible decrease in size compared with baseline), and (iii) no response / worsening (i.e., the BCC has not demonstrated any visible decrease in size compared with baseline).
Time Frame: Day 43
Population: Efficacy analysis set: the efficacy analysis set included all randomized participants with evaluable data.
Measure: Number; unit: Participants
Arm/Group | LDE225 0.75% | Vehicle
Number analyzed (Participants) | 16 | 8
Participants
  Complete response | 3 | 1
  Partial response | 9 | 4
  No response | 4 | 3

ADVERSE EVENTS:
Description: The nBCC participant from the LDE225 75% group was analyzed for safety as a separate arm.
Groups:
- LDE225 0.75% - sBCC: Participants topically applied 0.75% LDE225 cream twice daily for 6 weeks.
- Vehicle - sBCC: Participants topically applied matching placebo cream twice daily for 6 weeks.
Arm/Group | LDE225 0.75% - sBCC | Vehicle - sBCC | LDE225 0.75% - nBCC
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 8/16 | 5/8 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDE225 0.75% - sBCC (N=16) | Vehicle - sBCC (N=8) | LDE225 0.75% - nBCC (N=1)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gingival cyst (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Application site dermatitis (General disorders) | 0 | 1 | 0
Application site pruritus (General disorders) | 0 | 1 | 0
Local swelling (General disorders) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Application site folliculitis (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1
Glomerular filtration rate increased (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.